CLINICAL TRIAL: NCT03792451
Title: Nutrition Status of Adults With Phenylketonuria Treated With Pegvaliase
Brief Title: Nutrition Status of Adults Treated With Pegvaliase
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Krista Viau, Clinical Nutrition Specialist II, Boston Children's Hospital
Other Study IDs: P00029611
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pegvaliase — Treated with pegvaliase for one or more years or followed an unrestricted diet for 6 or more months while being treated with pegvaliase.
  Other Names: Palynziq

SUMMARY:
Conduct a cross-sectional analysis of the nutritional status of individuals with PKU treated with pegvaliase for one or more years or who have followed an unrestricted diet for 6 or more months while on pegvaliase treatment. We will evaluate laboratory markers of nutritional status, including markers of protein and micronutrient nutriture. In addition, a three-day food record and food frequency questionnaire will be obtained to assess protein intake and overall diet quality.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of phenylketonuria
2. Aged 18-65 years
3. Currently treated with pegvaliase
4. Have either 1) received treatment with pegvaliase for one or more years or 2) followed an unrestricted diet for 6 or more months while on pegvaliase
5. Currently following an unrestricted diet that meets or exceeds the RDA for protein (0.8 g/kg/day)

Exclusion Criteria:

1. Unable to consent to study
2. Under age 18 years or over age 65
3. Routine food intake provides less than the RDA for protein (0.8 g/kg/d)
4. Consuming any PKU medical foods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will recruit adults with PKU who have been treated with pegvaliase for one or more years or who have followed an unrestricted diet for 6 or more months while on pegvaliase treatment. This may include individuals who participated in the phase III clinical trials for pegvaliase.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mean concentrations of serum marker(s) of protein status | through study completion, an average of 1 year
Mean concentrations of serum marker(s) of micronutrient status | through study completion, an average of 1 year
Mean concentrations of serum marker(s) of essential fatty acid status | through study completion, an average of 1 year
Mean concentrations of serum marker(s) of cardiovascular status | through study completion, an average of 1 year
Mean protein intake (g/day) as reported on a three-day food record | through study completion, an average of 1 year
Mean micronutrient intake (%DRI) as reported on a three-day food record | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Mean Healthy Eating Index-2015 scores calculated from the Diet History Questionnaire III | through study completion, an average of 1 year
  "The Healthy Eating Index-2015 (HEI-2015) is… used to assess how well a set of foods aligns with the 2015-2020 Dietary Guidelines for Americans. The HEI-2015 includes 13 components that can be summed to a maximum total score of 100 points. The components capture… adequacy components and… moderation components. For the adequacy components, higher scores reflect higher intakes that meet or exceed the standards. For the moderation components, higher scores reflect lower intakes because lower intakes are more desirable. A higher total score indicates a diet that aligns better with the Dietary Guidelines." - https://www.cnpp.usda.gov/sites/default/files/healthy_eating_index/HEI2015-ScoresForAmericans.pdf
  Adequacy components include total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids. Moderation components include refined grains, sodium, added sugars, and saturated fats.
Correlation between serum micronutrient concentrations and average micronutrient intake | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Krista Viau, PhD, RD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No